CLINICAL TRIAL: NCT00726154
Title: Rhythmicity as a Moderator of Treatment Outcomes of Bipolar I Depression -Pilot Study
Brief Title: Pilot Study of the Effects of Circadian Rhythms on the Treatment of Bipolar I Depression.
Acronym: Rhythms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not receive funding
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 08020410
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Circadian Rhythm; Moderators; Lithium; Quetiapine
MeSH Terms: conditions — Bipolar Disorder | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPSRT (Other): Interpersonal and social rhythm therapy (IPSRT) focuses specifically on rhythmicity. IPSRT is based on the social zeitgeber hypothesis (Ehlers et al., 1988; 1993) and the conviction that regularity of social routines and stability of interpersonal relationships have a protective effect in recurrent mood disorders. In IPSRT, resolution of depressive symptoms is theorized to come about through the exploration of the links among mood symptoms, stability of social rhythms and quality of social relationships and social role performance, and the identification and management of potential precipitants of rhythm disruption.
  Interventions: Behavioral: IPSRT
- Collaborative care (Other): The collaborative care (CC) condition is a less intensive psychosocial intervention that was employed as the control condition in the STEP-BD study of psychosocial treatment (see Miklowitz et al., 2007). Participants assigned to this condition will receive a psychoeducational videotape and a workbook including information about: 1) the diagnosis, management, and treatment of bipolar illness; 2) the importance of medication adherence; 3) schedule management including daily mood charting; 4) typical biases in thinking relevant to mood states; 5) improving relationships through communication skills; and 6) developing a treatment contract geared toward preventing episodes.
  Interventions: Behavioral: Collaborative Care

INTERVENTIONS:
Behavioral: IPSRT — Interpersonal and social rhythm therapy (IPSRT) focuses specifically on rhythmicity. IPSRT is based on the social zeitgeber hypothesis (Ehlers et al., 1988; 1993) and the conviction that regularity of social routines and stability of interpersonal relationships have a protective effect in recurrent mood disorders. In IPSRT, resolution of depressive symptoms is theorized to come about through the exploration of the links among mood symptoms, stability of social rhythms and quality of social relationships and social role performance, and the identification and management of potential precipitants of rhythm disruption.
  Other Names: Psychotherapy
  Arms: IPSRT
Behavioral: Collaborative Care — The collaborative care (CC) condition is a less intensive psychosocial intervention that was employed as the control condition in the STEP-BD study of psychosocial treatment (see Miklowitz et al., 2007). Participants assigned to this condition will receive a psychoeducational videotape and a workbook including information about: 1) the diagnosis, management, and treatment of bipolar illness; 2) the importance of medication adherence; 3) schedule management including daily mood charting; 4) typical biases in thinking relevant to mood states; 5) improving relationships through communication skills; and 6) developing a treatment contract geared toward preventing episodes.
  Other Names: psychotherapy
  Arms: Collaborative care

SUMMARY:
The objective of this pilot study is to test the feasibility of a larger planned trial. The objective of this larger trial will be to determine the extent to which aspects of circadian rhythmicity, including, sleep/wake rhythms, daily social routines (i.e., social rhythms), circadian type (morningness/eveningness), endogenous circadian rhythms and polymorphisms associated with altered circadian function in specific genes (namely, CLOCK, Period 2 and Period 3) moderate treatment response in bipolar disorder.

DETAILED DESCRIPTION:
This study is a small scale pilot study which will be used to support a larger trial. The major aims of the larger study are to determine the extent to which aspects of circadian rhythmicity, including, sleep/wake rhythms, daily social routines (i.e., social rhythms), circadian type (morningness/eveningness), endogenous circadian rhythms and polymorphisms associated with altered circadian function in specific genes (namely, CLOCK, Period 2 and Period 3) moderate treatment response in bipolar disorder.

The overarching aim of the study is to clarify the nature of rhythm abnormalities in bipolar disorder and, especially, their relation to clinical state. We propose to do this in the context of a randomized intervention protocol in which half of the subjects will receive a treatment aimed at rhythm regularization. We expect to study individuals with a range of circadian and sleep-wake abnormalities, social rhythm disturbances, and circadian type and to examine the extent to which these parameters predict subjects' clinical outcomes. Since one half of the subjects will receive IPSRT as part of their treatment regimen (with increasing regularity of social routines as a goal of treatment), we will be able to examine the extent to which changes in social rhythm regularity and sleep quality are associated with clinical and functional improvement and whether these outcomes are mediated by changes in endogenous circadian rhythms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years
2. Able to give basic informed consent
3. Meets DSM-IV criteria for current acute episode of bipolar I depression
4. Women of childbearing potential must agree to use a doctor-approved birth control throughout participation in the study
5. Hamilton Depression Rating Scale (17-item) score > or equal to 15
6. Hamilton Depression Rating Scale (17-item) item 1 score > or equal to 2
7. Young Mania Rating Scale score < or equal to 12

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements (i.e., complete forms, attend scheduled evaluations)
2. Not competent to provide informed consent in the opinion of the investigator
3. Rapid cycling (4 or more episodes per year) bipolar I disorder
4. Present treatment for index depressive episode with lithium or quetiapine unless does or serum level are deemed inadequate
5. Lithium intolerance or a past failed adequate trial of Lithium
6. Quetiapine intolerance or a past failed adequate trial of quetiapine
7. Presence of schizophrenia, schizoaffective, antisocial or pervasive developmental disorder, psychotic disorder, current substance dependence, and organic mental disorder
8. Axis II borderline disorder
9. Mini-Mental State Examination score <24
10. Current alcohol and illicit substance abuse
11. Women who are currently pregnant, planning to become pregnant or currently breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
This is a pilot feasibility study. The primary endpoint is depression severity at week 16, which will be measured via the Hamilton Rating Scale for Depression 25-item score (HRSD-25). | 2 years

SECONDARY OUTCOMES:
Other secondary endpoints include the social rhythm regularity, sleep/wake function, quality of life, social and occupational functioning. These will be measured by various data collection forms and questionnaires | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States